CLINICAL TRIAL: NCT05428904
Title: Developing a Virtual Reality-Based Simulation Program for Nursing Students and Using in Nursing Research
Brief Title: Virtual Reality Simulation for Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe ARIKAN DÖNMEZ, Asst. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KA-21126
Record Dates: First submitted 2022-04-13; First posted 2022-06-23 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Nursing Education; Virtual Reality; Simulation; Satisfaction; Critical Thinking
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Nursing undergraduate students participating in a virtual reality simulation program
  Interventions: Other: Virtual Reality Simulation
- Control Group (No Intervention): Nursing undergraduate students receiving attention-matched training

INTERVENTIONS:
Other: Virtual Reality Simulation — Virtual reality applications are a type of three-dimensional computer-based simulation that gives a sense of being anywhere and provides various data to the sense organs for this. However, virtual reality applications are a simulation model that creates a sense of reality for the participants and allows mutual communication with a computer-based dynamic environment.
  Arms: Intervention Group

SUMMARY:
Today, thanks to the developing hardware technology, various distance education projects are carried out with virtual reality, augmented reality and even mixed reality glasses. The visual writing fields of the content they provide can be extended as much as necessary.

With this research, it is aimed to develop a virtual reality-based simulation program and to ensure its use in nursing education and research.

DETAILED DESCRIPTION:
The universe of the research will consist of 219 students who are studying at Hacettepe University Faculty of Nursing in the Spring Semester of the 2021-2022 Academic Year and who have successfully completed the Internal Medicine Nursing course. As a result of the power analysis, it is aimed to reach a total of 100 people, with 50 students in each group. Our research was planned in a randomized controlled design. The data of the research will be collected through Student Information Form, Knowledge Tests, Perceived Learning Scale, General Self-Efficacy Scale, Satisfaction with Educational Methods Questionnaire and California Critical Thinking Disposition Scale. With this research, it is predicted that there will be an increase in nursing students' knowledge score, perceived learning, general self-efficacy, satisfaction with the education method, and critical thinking dispositions.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completing the Internal Medicine Nursing Course
* Having internet access
* Volunteering to participate in the research

Exclusion Criteria:

* Not being able to communicate in Turkish
* Being in the intervention groups and not participating in the virtual simulation application
* Not participating in any of the pre-test, post-test, or follow-up tests

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Knowledge Tests | Changes from baseline to one day post-test and after one month follow-up
  In order to determine the cognitive learning of the students, questionnaires consisting of 20 multiple-choice questions for each subject and to be evaluated over 100 points will be created. A literature review will be made for the creation of questionnaires and these forms will be created to determine cognitive competencies in line with the educational content. Validity and reliability studies will be conducted to test the usability of the forms.
Perceived Learning Scale | Changes from baseline to one day post-test and after one month follow-up
  Perceived Learning Scale Rovai et al. (2009) developed by. The validity and reliability studies of the scale were performed by Albayrak et al. (2004) with 227 university students. The scale has 9 items and three factors, and the first factor is "Cognitive", which includes three items aiming to measure cognitively perceived learning. The second factor was named "Affective", which includes three items aiming to measure learning perceived as affective, and the third factor, "Psychomotor", which aims to measure learning perceived as psychomotor. A score between 9 and 63 is obtained from the entire scale. An increase in the scale score indicates an increase in the perceived learning level. The Cronbach's alpha, which includes all nine items of the scale for internal consistency, was .83.
Satisfaction Survey with Training Methods | Changes from baseline to one day post-test and after one month follow-up
  Training methods satisfaction questionnaire was developed by Gürpınar (Cronbach alpha: 0.84) and used in his studies. The questionnaire consists of 16 propositions. One of these propositions is the proposition "I am satisfied with this education method in general", which questions the state of being satisfied with the education. Other propositions were formed from propositions aiming to determine the views of the education method in general about the contribution of the education method to the learning and professional life of the student. It is determined that as the scale score average increases, the satisfaction of the students in the education method increases, and as the scale score average decreases, their satisfaction in the education method decreases. In the evaluation of the scale, students are given a minimum of 16 and a maximum of 80 points for their satisfaction with education methods. Atan et al. (2019), the Cronbach alpha value of the scale was found to be 0.90.
Critical Thinking Disposition Scale | Changes from baseline to one day post-test and after one month follow-up
  This scale was developed by Facione in 1990, and its validity and reliability study in Turkey was carried out by Kökdemir in 2003. It consists of 51 items and six subscales. The scale is a six-item Likert-type scale. The score range of the scale is 51-306. A low score indicates a low critical thinking disposition, and a high score indicates a high critical thinking disposition. The Cronbach's alpha value of the scale was found to be 0.88.
General Self-Efficacy Scale | Changes from baseline to one day post-test and after one month follow-up
  The Turkish validity and reliability study of the General Self-Efficacy scale, which was developed by Schwarzer and Jarusalem in Germany in 1981, was performed by Aypay (2010). The scale, which is all positive and consists of 10 items, was prepared in a 4-point Likert type limited to completely wrong and completely true points. All items are positively scored and a score between 10 and 40 is obtained. A high score means high general self-efficacy. The cronbach's alpha coefficient of the scale was found to be 0.83.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No